CLINICAL TRIAL: NCT07191444
Title: Efficacy and Safety of Firsekibart Versus Anakinra in Adult-Onset Still's Disease
Brief Title: A Study of Firsekibart Versus Anakinra in Adult-Onset Still's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IMM-M-L-002
Record Dates: First submitted 2025-09-01; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-08

CONDITIONS: Still's Disease, Adult-Onset
MeSH Terms: interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Firsekibart group
  Interventions: Biological: Firsekibart
- Anakinra group
  Interventions: Biological: Anakinra

INTERVENTIONS:
Biological: Firsekibart — Firsekibart will be administered according to the protocol
  Groups: Firsekibart group
Biological: Anakinra — Anakinra will be administered according to the protocol
  Groups: Anakinra group

SUMMARY:
The purpose of this study is to compare the efficacy and safety of firsekibart versus anakinra in patients with AOSD.

ELIGIBILITY:
Inclusion Criteria:

* Age: This study will include subjects aged 18 to 75 years (inclusive), regardless of gender.
* Subjects must be willing to participate in the study and voluntarily sign an informed consent form.
* Diagnosis of AOSD will be based on the Yamaguchi criteria: Major criteria: (1) Fever ≥39°C lasting for ≥1 week; (2) Arthralgia lasting for ≥2 weeks; (3) Typical rash; (4) White blood cell count ≥10×10^9/L with neutrophils ≥80%. Minor criteria: (1) Sore throat or pharyngitis; (2) Lymphadenopathy and/or splenomegaly; (3) Abnormal liver function; (4) Negative rheumatoid factor and antinuclear antibody. Exclusion criteria: (1) Infectious diseases (especially sepsis and EBV infection); (2) Malignancies (especially lymphoma); (3) Other rheumatic diseases (particularly systemic vasculitis). After excluding the above exclusion criteria, a diagnosis of AOSD requires meeting ≥5 of the above criteria (including at least 2 major criteria).
* Active disease is defined as meeting 2 Yamaguchi criteria along with the presence of fever or CRP >10 mg/L.
* If currently receiving glucocorticoid therapy, the dose must have been stable for at least 1 week prior to randomization. The maximum allowed dose is 1 mg/kg/day.
* Subjects (including their partners) must have no pregnancy plans from the screening period until 28 days after the last dose and must voluntarily use contraception.

Exclusion Criteria:

* Pre-randomization Medications: a) Received BTK inhibitors, JAK inhibitors, intravenous immunoglobulin, plasmapheresis, or traditional Chinese medicine within 4 weeks prior to screening or 5 half-lives of the known drug (whichever is shorter). b) Received anakinra therapy within 1 day prior to randomization. c) Received etoposide (VP-16) therapy within 12 weeks prior to the baseline visit. d) Increase in dose or addition of new non-biologic agents for treating rheumatic/autoimmune diseases (e.g., immunosuppressants, immunomodulators, antimalarials) within 3 days prior to the baseline visit, unless deemed ineffective by the investigator and discontinued prior to baseline. Specific agents include: i Immunosuppressants/Immunomodulators: Methotrexate, azathioprine, leflunomide, mycophenolate mofetil (or mycophenolate sodium), mizoribine, calcineurin inhibitors (e.g., tacrolimus, cyclosporine), sirolimus, oral cyclophosphamide, 6-mercaptopurine, thalidomide, total glucosides of paeony. ii Antimalarials: Hydroxychloroquine, chloroquine, quinacrine.
* History of hypersensitivity to any component of the investigational product.
* Presence or suspicion of hemophagocytic lymphohistiocytosis (HLH) at baseline, or diagnosis of HLH within 2 months prior to randomization. According to the HLH-2004 diagnostic criteria, the diagnosis can be established by meeting any one of the following two conditions: (1) Molecular diagnosis consistent with HLH. (2) Fulfillment of ≥5 of the following 8 criteria: a) Fever: Temperature >38.5°C for >7 days. b) Splenomegaly. c) Cytopenias (affecting ≥2 lineages): Hemoglobin <90 g/L, neutrophils <1.0×10⁹/L, not due to reduced bone marrow function. d) Hypertriglyceridemia and/or hypofibrinogenemia: Triglycerides ≥ 3 mmol/L or >3 SD above age-specific norms, and/or Fibrinogen ≤ 1.5 g/L or <3 SD below age-specific norms.e) Identification of hemophagocytes in bone marrow, spleen, or lymph nodes. f) Elevated serum ferritin (≥500 μg/L). g) Low or absent NK cell activity. h) Elevated soluble IL-2 receptor (sCD25 ≥2400 U/mL).
* Hematologic Diseases: History or current presence of hematologic disorders (including but not limited to myelofibrosis, aplastic anemia, leukemia, lymphoma).
* Cardiovascular Diseases: Acute myocardial infarction or unstable angina within 6 months; severe arrhythmias (multifocal frequent ventricular premature beats, ventricular tachycardia, ventricular fibrillation); NYHA Class III-IV heart failure.
* Pulmonary Diseases: Including but not limited to asthma, COPD, interstitial lung disease, pulmonary alveolar proteinosis, or pulmonary granulomatosis, with abnormal pulmonary function tests (FVC <80% predicted or FEV1/FVC <70%); or any pulmonary condition deemed by the investigator to significantly impair lung function and unsuitable for study participation.
* Malignancy: History of malignancy within the past 5 years (regardless of treatment), except successfully treated basal cell or squamous cell skin carcinoma.
* Other Diseases: Current clinically significant, unstable, or inadequately controlled acute/chronic diseases (e.g., acute pneumonia, pulmonary hypertension, diabetic ketoacidosis, acute pancreatitis); or planned medical/surgical procedures that may place the subject at undue risk or impair their ability to participate.
* Mycobacterium tuberculosis infection, including latent infection with positive T-SPOT.TB or PPD test.
* Positive serology for HBsAg, HBcAb, HCV-Ab, HIV-Ab, or Treponema pallidum antibody (by TPPA). If HBcAb is positive, HBV-DNA must be below the lower limit of quantification.
* Infection: Uncontrolled infection at screening as judged by the investigator (e.g., tuberculosis, pneumocystis, cytomegalovirus, herpes simplex, herpes zoster, atypical mycobacteria, Histoplasma capsulatum, Salmonella; or recurrent sinusitis, genital herpes, osteomyelitis, urinary tract infections).
* Surgery/Other Conditions: Planned surgery or any other medical history, laboratory abnormality, or condition that, in the investigator's judgment, renders the subject unsuitable for the study.
* Transplant History: History of major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplant.
* Renal impairment: Serum creatinine or BUN >1.5 × ULN; or eGFR ≤60 mL/min/1.73m² (calculated by MDRD formula: eGFR = 186 × [SCr (mg/dL)]-¹.¹⁵⁴ × [Age]-⁰.²⁰³ × [0.742 if female] × 1.233) prior to screening.
* Pregnancy or lactation.
* Participation in any clinical trial (including investigational vaccines) within 3 months prior to enrollment, or previous use of invasive investigational medical devices, or current enrollment in an interventional study.
* Live vaccination within 30 days prior to screening.
* History or evidence of alcohol abuse within 3 months prior to screening.
* Positive urine drug screen for morphine, ketamine, tetrahydrocannabinol, methamphetamine, or methylenedioxymethamphetamine.
* Any other condition that, in the investigator's opinion, would increase the risk associated with study participation, interfere with the evaluation of the investigational product, or confound the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study participants will be patients with active Adult-Onset Still's Disease recruited from Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-18 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects achieving clinical inactive disease (CID) at Week 24, where CID is defined as the absence of Still's disease-related symptoms with normal ESR or CRP levels. | At Week 24 from initiation of treatment

SECONDARY OUTCOMES:
Proportion of subjects achieving afebrile status with either ≥50% reduction in CRP levels or CRP within normal range at Weeks 2, 4, and 8. | At Weeks 2, 4, and 8 after treatment initiation
  Efficacy Endpoints
Proportion of subjects achieving afebrile status with either ≥70% reduction in CRP levels or CRP within normal range at Week 12. | At Week 12 after treatment initiation
  Efficacy Endpoints
Proportion of subjects achieving afebrile status with either ≥70% reduction in CRP levels or CRP within normal range, and glucocorticoid dose ≤0.2 mg/kg/day at Week 12. | At Week 12 after treatment initiation
  Efficacy Endpoints
Proportion of subjects achieving afebrile status with either ≥70% reduction in CRP levels or CRP within normal range, and glucocorticoid dose ≤0.1 mg/kg/day at Week 12. | At Week 12 after treatment initiation
  Efficacy Endpoints
Proportion of subjects achieving clinical inactive disease (CID) with discontinuation of glucocorticoids | At Week 24 after treatment initiation
  Efficacy Endpoints
Proportion of subjects without disease relapse at Weeks 12 and 24. | At Weeks 12 and 24 after treatment initiation
  Efficacy Endpoints
ACR30, ACR50, ACR70, and ACR90 response rates at Weeks 2, 4, 8, 12, 16, 20, and 24. | At Weeks 2, 4, 8, 12, 16, 20, and 24 after treatment initiation
  Efficacy Endpoints
Change from baseline in ferritin levels at Weeks 2, 4, 8, 12, 16, 20, and 24. | At Weeks 2, 4, 8, 12, 16, 20, and 24 after treatment initiation
  Efficacy Endpoints
Change from baseline in cytokine levels (including sIL-2R) at Weeks 2, 4, 8, 12, 16, 20, and 24. | At Weeks 2, 4, 8, 12, 16, 20, and 24 after treatment initiation
  Efficacy Endpoints
Change from baseline in ESR at Weeks 2, 4, 8, 12, 16, 20, and 24. | At Weeks 2, 4, 8, 12, 16, 20, and 24 after treatment initiation
  Efficacy Endpoints
Change from baseline in CRP levels at Weeks 2, 4, 8, 12, 16, 20, and 24 | At Weeks 2, 4, 8, 12, 16, 20, and 24 after treatment initiation
  Efficacy Endpoints
Change from baseline in Pouchot score at Weeks 2, 4, 8, 12, 16, 20, and 24. | At Weeks 2, 4, 8, 12, 16, 20, and 24 after treatment initiation
  Efficacy Endpoints. Pouchot score ranges from 0 to 12 points, with higher scores indicating a poorer outcome.
Change from baseline in glucocorticoid dose at Weeks 2, 4, 8, 12, 16, 20, and 24. | At Weeks 2, 4, 8, 12, 16, 20, and 24 after treatment initiation
  Efficacy Endpoints
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: No